CLINICAL TRIAL: NCT04980651
Title: Safety and Efficacy of Remote Ischemic Conditioning for Acute Ischemic Stroke: A Multicenter, Randomized, Parallel-controlled Clinical Trial
Brief Title: Safety and Efficacy of Remote Ischemic Conditioning for Acute Ischemic Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yi Yang (Other)
Responsible Party: Sponsor-Investigator, Yi Yang, Associated Dean of First Hospital of Jilin University, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SERIC
Record Dates: First submitted 2021-07-13; First posted 2021-07-28 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-02

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIC+Standard medical treatment (Active Comparator): Remote ischemic conditioning (RIC) is induced by 4 cycles of 5 min of healthy upper limb ischemia followed by 5 min reperfusion. Limb ischemia was induced by inflation of a blood pressure cuff to 200 mm Hg. RIC will be conducted twice daily for 7 consecutive days. Additionally, the patients will be treated with standard medical treatment according to the Guidelines for diagnosis and treatment of acute ischemic stroke in China 2014.
  Interventions: Procedure: Remote ischemic conditioning
- Sham RIC+Standard medical treatment (Placebo Comparator): Remote ischemic conditioning (RIC) is induced by 4 cycles of 5 min of healthy upper limb ischemia followed by 5 min reperfusion. Limb ischemia was induced by inflation of a blood pressure cuff to 60 mm Hg. RIC will be conducted twice daily for 7 consecutive days. Additionally, the patients will be treated with standard medical treatment according to the Guidelines for diagnosis and treatment of acute ischemic stroke in China 2014.
  Interventions: Procedure: Sham remote ischemic conditioning

INTERVENTIONS:
Procedure: Remote ischemic conditioning — Remote ischemic conditioning (RIC) is induced by 4 cycles of 5 min of healthy upper limb ischemia followed by 5 min reperfusion. Limb ischemia was induced by inflation of a blood pressure cuff to 200 mm Hg.
  Arms: RIC+Standard medical treatment
Procedure: Sham remote ischemic conditioning — Sham remote ischemic conditioning (RIC) is induced by 4 cycles of 5 min of healthy upper limb ischemia followed by 5 min reperfusion. Limb ischemia was induced by inflation of a blood pressure cuff to 60 mm Hg.
  Arms: Sham RIC+Standard medical treatment

SUMMARY:
The purpose of this study is to determine the efficacy and safety of remote ischemic conditioning for acute ischemic stroke.

DETAILED DESCRIPTION:
In this study, 2210 cases of ischemic stroke in 72 hours were included in 10 centers in China according to the principle of random, and parallel control. The experimental group receive basic treatment and remote ischemic conditioning for 200mmHg, 2 times per day for 7 consecutive days. The control group receive basic treatment and remote ischemic conditioning control for 60mmHg, 2 times per day for 7 consecutive days. Two groups will be followed up for 90 days to evaluate the efficacy and safety of remote ischemic conditioning in treating acute ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* 1) Age≥18 years, regardless of sex.
* 2) Patients with clinically definite diagnosis of acute ischemic stroke and able to commence RIC treatment within 72 hours of stroke onset.
* 3) Baseline NIHSS ≥ 4, ≤ 24.
* 4) Baseline mRS ≤ 2;
* 5) Signed and dated informed consent is obtained.

Exclusion Criteria:

* 1) Patients who undergo thrombolytic therapy or endovascular treatment.
* 2) The patients who had the contraindication of remote ischemic conditioning treatment, such as severe soft tissue injury, fracture, or vascular injury in the upper limb. Acute or subacute venous thrombosis, arterial occlusive disease, subclavian steal syndrome, etc.
* 3) Other intracranial lesions, such as cerebrovascular malformation cerebral venous diseases, tumors,s and other diseases involving the brain.
* 4) Pregnant or lactating women.
* 5) Previous remote ischemic conditioning therapy or similar treatment.
* 6) Severe hepatic and renal dysfunction.
* 7) Patients with a life expectancy of less than 3 months or patients unable to complete the study for other reasons.
* 8) Unwilling to be followed up or treated for poor compliance.
* 9) He/She is participating in other clinical research or has participated in other clinical research or has participated in this study within 3 months prior to admission.
* 10) Other conditions that the researchers think are not suitable for the group.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2210 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with modified Rankin Scale (mRS) Score 0-2. | 3 months
  Proportion of patients with modified Rankin Scale (mRS) Score 0-2. Ranged from 0 to 6, a low value represents a better outcome.

SECONDARY OUTCOMES:
National Institute of Health stroke scale (NIHSS) at 7 days, 30±3 days, 90±3 days from onset. | 7days, 30±3 days, 90±3 days
  National Institute of Health stroke scale (NIHSS) at 24 hours, 7 days, 30±3 days, 90±3 days from onset. Ranged from 0 to 42, a low value represents a better outcome.
modified Rankin Scale (mRS) Score at 7 days, 30±3 days, 90±3 days from onset. | 7days, 30±3 days, 90±3 days
  modified Rankin Scale (mRS) at 24 hours, 7 days, 30±3 days, 90±3 days from onset. Ranged from 0 to 6, a low value represents a better outcome.
Barthel Index (BI) at 7 days, 30±3 days, 90±3 days from onset. | 7days, 30±3 days, 90±3 days
  Barthel Index (BI) at 7 days, 30±3 days, 90±3 days from onset. Ranged from 0 to 100, a high value represents a better outcome.
Proportion of patients with hemorrhagic transformation during hospitalization. | 7 days
  Proportion of patients with hemorrhagic transformation during hospitalization.
Frequency of adverse events during follow-up. | 90 days
  Severe adverse events through day-90 after the onset of acute ischemic stroke.

OTHER OUTCOMES:
Blood pressure at 24 hours, 7 days, 30±3 days, 90±3 days. | 24 hours, 7 days, 30±3 days, 90±3 days
  Blood pressure at 24 hours, 7 days, 30±3 days, 90±3 days.
heart rate at 24 hours, 7 days, 30±3 days, 90±3 days. | 24 hours, 7 days, 30±3 days, 90±3 days
  heart rate at 24 hours, 7 days, 30±3 days, 90±3 days.
Numeric rating scales (NRS) score during intervention. | 7 days
  Numeric rating scales (NRS) score during intervention. Ranged from 0 to 10, a low value represents a less pain.
Proportion of patients with early withdrawal for safety or tolerability reasons. | 7 days
  Proportion of patients with early withdrawal for safety or tolerability reasons.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China